CLINICAL TRIAL: NCT03971448
Title: Randomized Control Trial of Casting Versus Pediatric Walker-Boot in the Management of Toddler's Fractures
Brief Title: Toddlers Fractures - Cast Versus Removable Boot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Population Services International (Other)
Responsible Party: Principal Investigator, Kathy Boutis, Staff Emergency Physician, Research and PRAISE Director, Sr. Associate Scientist, Child Health Evaluative Sciences, Research Institute, The Hospital for Sick Children, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000063960
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Toddler's Fracture
Keywords: Cast; Removable device/boot; Immobilization strategy; Emergency Department
MeSH Terms: conditions — Tibial Fractures; Emergencies

STUDY DESIGN:
Intervention Model Description: Enrolled children will be randomly assigned to either a fiberglass above-knee walking cast (AKWC) or the Landmark Pediatric Walker Boot (LPWB).
Who Masked: Outcomes Assessor
Masking Description: Double blinding is not feasible since the patient and families will know which immobilization method was applied. Therefore, the individual performing the outcome assessments will be a different person from the research team and will be masked to treatment allocation. The families will be instructed not to reveal the allocation to the research team member in order to minimize the chances of unblinding during follow-up encounters. In spite of the latter, there is potential for accidental unblinding. The frequency of this will be documented and reported.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiberglass above-knee walking cast (AKWC) (Active Comparator): The standard treatment arm will be a posterior splint placed in the ED by the ED clinical team (nurse/physician) and then a fiberglass AKWC to be placed ideally within 72 hours in the fracture clinic. This AKWC will be in place for 3 weeks, which is currently the most common strategy to manage TF.
  Interventions: Device: AKWC
- Landmark Pediatric Walker Boot (LPWB) (Experimental): The Landmark Pediatric Walker Boot (LPWB) will be placed in the ED and will be kept on for a minimum of one week, and then for a duration dictated by the patient's comfort.
  Interventions: Device: LPWB

INTERVENTIONS:
Device: LPWB — The LPWB will be placed by clinical staff who will have been trained on the proper application of this device at the initial ED visit. At ED discharge, both populations will receive identical documentation on recommendations for weight bearing, type and frequency of analgesics, reasons to return for medical attention. The only difference will be care instructions related to the specific immobilization device. Specifically, the experimental group will be permitted to remove the LPWB as early as one week post ED visit as tolerated by the patient's symptoms.
  Arms: Landmark Pediatric Walker Boot (LPWB)
Device: AKWC — If the patient is randomised to AKWC, it will be apply by a cast technician. Children with AKWC immobilization will be provided with up to two appointments in the orthopedic clinic. In case the AKWC could not been placed at initial visit, the first will be within 72 hours of the ED visit to have the fiberglass AKWC placed. The second appointment will be for cast removal.
  Arms: Fiberglass above-knee walking cast (AKWC)

SUMMARY:
A toddler's fracture is a fracture that occurs in the lower leg, oven the shin, of children 9 months to four years of age. It usually happens when a young child twists the leg while running or jumping. It is one of the most common injuries of the leg in this age group. In Canada and the United States there are about 80,000 cases per year that present to emergency departments. The good news is that these fractures are stable injuries and heal exceptionally well, without any reported concerns for problems in the future. Despite this, most children with this fracture are managed in a restrictive full circular cast, often including the entire leg, for three to six weeks. This cast management then also includes about two to three repeat visits to see a bone doctor, where the cast is often changed and new x-rays are taken with each visit. However, none of these things has ever been shown to change the way these young children's fractures heal. Further, casting can cause harm such as skin irritation or poor cast fit which may result in problems that are more distressing than the fracture itself. There are also costs to consider. The needless excess costs of the current management strategy in Canada alone can be estimated to be about 1.8 million dollars annually. And so, increasingly, some doctors are choosing to manage these stable fractures with a supportive device on the lower leg, a removable walking boot. This type of device can be taken off as needed by the parent and child and used only as long as the child needs it to manage the pain that results from this stable fracture. This makes caring for the child much easier and allows the child to return to activities when the child is ready. Further, families do not necessarily need to return to a bone doctor for cast changes or x-rays or reassessment. Since this fracture recovers so well, patients can see their family doctor to make sure their child is returning to activity as expected and have their questions about recovery answered. But, in order to be sure that the removable walking boot works as well as a cast in these fractures, we need to do a well-designed study to make sure we consider all the important aspects of making this change. As a result, in children with toddler's fractures, we will compare the traditional treatment of cast placement to a removable walking boot with respect to how each immobilization strategy controls pain and how quickly children return to their usual activities. We hope that children treated with a removable walking boot will still be able to achieve good pain control while their injury is healing. It is possible too those children will even return to their activities sooner and this newer strategy could save the health care system money.

DETAILED DESCRIPTION:
Background:

Toddler's fractures (TF) are characterized as stable, spiral or oblique fractures of the tibial diaphysis or distal metaphysis that mainly occur in children between nine months and four years of age. Despite its inherent stability, the most frequent treatment option remains an above/below knee casting for three to six weeks, without clear and strong evidence to do so. Casting and orthopedic follow-up results in further burden including unnecessary visits to an orthopedic surgeon, additional sets of lower extremity radiographs and day-to-day inconveniences/complications (e.g. bathing/showering, problems of fit, breakage, and skin related complications). Commercially available removable immobilization devices have been applied successfully to low-risk stable extremity pediatric fractures, and have numerous advantages over conventional immobilization with casts (e.g. easy care, comfort and application/removal convenience) but have not properly been studied in the management of TF.

Study Aims:

To compare the recovery of children with TF when treated with a commercial, removable immobilization device versus an above-knee walking fiberglass cast.

Hypothesis:

The removable pediatric walking boot will be at least as effective as the walking above-knee cast with respect to pain with ambulation as measured by the EVENDOL scale at four weeks after injury.

Research Design:

This is a multi-centre, two-arm, non-inferiority randomized control trial. All independently weight-bearing children age 9 months to 4 years who present to the ED within five days of a lower extremity injury/complaint and diagnosed clinically and radiolographically with an accidental TF will be eligible for enrolment. Study participants will be randomly assigned to receive either a removable below knee device or a circumferential walking cast. The main outcome will be pain with ambulation as measured by the EVENDOL pain scale at four weeks. Complications, day-to-day burdens, unscheduled visits will be ascertained, as the impact and satisfaction with the treatment device. Accounting to a maximal 20% drop-off rate, a sample size of 160 participants was calculated to have a power of 90% to identify a difference of 2 with an alpha value of 0.025. About one-third of participants will be recruited at CHU Sainte-Justine (n=54).

Relevance:

Current practice patterns predominately include treatment with a circumferential cast for several weeks. This type of rigid immobilization is likely unnecessary for such a stable injury. However, the research to date comparing casting with removable devices in children with TF has significant limitations and has not been of sufficient quality to change the immobilization and follow-up practice of TF. Specifically, retrospective design and analyses of data collected for a different purpose is subject to methodological limitations such as bias, missing data, and inconsistent measurement of outcomes. Further, these data have typically been limited to a single site, limiting generalizability. Other research has gathered data using surveys, which is limited by the fact that what physicians say they do does not necessarily represent what they actually do, and hence does not necessarily accurately represent clinical practice or outcomes. Finally, no research to date has considered the perspectives of families who need to care for these injured toddlers at home. Therefore, to secure the confidence of all relevant stakeholders, we need to provide high quality evidence to determine the most effective and convenient management strategy for this common childhood injury. If we can demonstrate that a removable device is at least as safe and effective as a circumferential cast in the treatment of TF, there are likely to be similar benefits for these fractures as it has been found with other minor pediatric fractures (e.g. comfort/convenience, safety, recovery, and cost-effectiveness advantages). As this is a common injury in childhood, the use of a removable device to manage this injury is highly likely to result in lower morbidity and save costs for the health care system and population, and these advantages will also generalize nationally and internationally.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy, independently weight-bearing children aged 9 months to 4 years
* Present to the ED at SickKids, LHSC or CHU Sainte-Justine within five days of a lower extremity injury
* Diagnosed clinically and radiographically with an accidental TF will be eligible for enrolment

Exclusion Criteria:

* Children at risk for pathological fractures (Appendix 1) or those with chronic conditions (arthritis or neuromuscular disorders) since these children have different management requirements and potentially different pain and recovery timelines
* Children with multi-limb injuries
* Children with neuromotor deficits such that assessment of recovery or pain is confounded by the deficits
* Children whose parents/guardians who are unable to provide consent or complete follow-up procedures due to an insurmountable language barrier, or no access to a phone or electronic mail
* Children with diagnostic uncertainty of a TF (e.g. occult TF) or those whose TF might be the result of non-accidental injury

Ages: 9 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
EValuation ENfant DOuLeur (EVENDOL) pain score at four weeks | 4 weeks post injury
  In this scale, there are five items (scored 0 to 3) using two simultaneous criteria (intensity and duration of the behaviour) for a total score that ranges from 0 to 15. Using this measurement, higher scores indicate more pain, and a score of at least four should trigger a clinician to provide pharmacological analgesia.

SECONDARY OUTCOMES:
Complications | 4 and 12 weeks post injury
  Proportion of complications within four weeks post index ED visit. Complications will be a composite outcome of any of the following: pain, skin irritation, infection, immobilization device fitting issues or breakage, thermal injury, cast saw injury, and protracted limping.
Weight-bearing as per baseline | 2, 4 and 12 weeks post-injury
  Proportion of children that weight bear as per pre-injury baseline "most of the time"
Unscheduled visits | 4 weeks post injury
  Proportion of children with unscheduled visits to a physician for the index injury, measured by parental report and Canadian Institute of Health Information data.
Day-to-day issues | 4 weeks post injury
  Parental perceptions of challenging issues during the four weeks post-injury will be measured using a five point Likert Scale
Immobilization strategy satisfaction | 4 weeks post injury
  Proportion of parents who were at least "satisfied" with the treatment device measured on a five point Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Plan for future analyses and would need a data sharing agreement.

REFERENCES:
- [Derived] Boutin A, Colaco K, Stimec J, Camp M, Narayanan U, Bhatt M, Poonai N, Willan AR, Cook R, Nault ML, Carsen S, Boutis K. Removable Boot vs Casting of Toddler's Fractures: A Randomized Clinical Trial. JAMA Pediatr. 2025 Apr 21;179(7):713-21. doi: 10.1001/jamapediatrics.2025.0560. Online ahead of print. PMID 40257790